CLINICAL TRIAL: NCT05826795
Title: Cost-effectiveness of Applying Early Goal-directed Therapy Using FloTrac/EV1000 Platform in Patients Undergoing Coronary Artery Bypass Graft With Cardiopulmonary Bypass
Brief Title: Cost-effectiveness of EGDT Using FloTrac/EV1000
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Other Study IDs: HE631648
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease
Keywords: Cost-effectiveness; Early goal-directed therapy; FloTrac/EV1000; ICU stay
MeSH Terms: conditions — Coronary Artery Disease | interventions — Early Goal-Directed Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: During the intraoperative period, both before and after CPB, the Control group received fluid, inotropic, and/or vasoactive drugs at the discretion of the attending anesthesiologists to achieve the following goals: MAP 65-90 mmHg; CVP 8-12 mmHg; urine output ≥ 0.5 mL·kg-1·h-1; SpO2 > 95%; and hematocrit 26-30%. Arterial blood gas (ABG) and electrolytes were monitored and corrected hourly.
- EV1000: The patients were managed to achieve similar goals: MAP 65-90 mmHg; urine output ≥ 0.5 mL·kg-1·h-1; SpO2 > 95%; and hematocrit 26-30%, using information from the FloTrac/EV1000. The EGDT group received: fluid to maintain a SVV < 13%; inotropic drugs to achieve a SVI of 33-65 mL·beat-1·m-2 and CI of 2.2-4.0 L·min-1·m-2; and/or vasoactive drugs to achieve a SVRI of 1600-2500 dynes·s·cm-5·m-2. ABG and electrolytes were monitored and corrected in the same manner.
  Interventions: Procedure: Early goal-directed therapy (EGDT)

INTERVENTIONS:
Procedure: Early goal-directed therapy (EGDT) — The principle of hemodynamic optimization to achieve the defined goals.
  Other Names: FloTrac/EV1000 platform
  Groups: EV1000

SUMMARY:
Coronary artery bypass graft (CABG) with cardiopulmonary bypass (CPB) is a high-risk surgery with significant morbidity that results in a prolonged stay in the intensive care unit (ICU) at an increased cost. Early goal-directed therapy (EGDT) using the FloTrac/EV1000 platform improved outcomes in these patients with shorter ICU stay but with extra cost for a FloTrac transducer. The objective of this study is to assess the cost-effectiveness of implementing the FloTrac/EV1000 in these patients.

DETAILED DESCRIPTION:
EGDT using FloTrac/EV1000 platform has been reported to improve outcomes in patients undergoing CABG with CPB resulting in a reduction in cardiovascular and thoracic ICU (CVT ICU) and hospital stay. However, the use of the FloTrac sensor has an extra cost that impedes its implementation. There is still no study that assesses the cost-effectiveness of implementing FloTrac in cardiac surgery.

The objective of our study is to evaluate the cost-effectiveness of applying EGDT using the FloTrac/EV1000 platform in patients undergoing CABG with CPB.

There are 2 steps in this study:

1. Assessing the efficacy of the FloTrac/EV1000 platform
2. Assessing the daily CVT ICU cost

Assessing the efficacy of the FloTrac/EV1000 platform

We compare the efficacy of the FloTrac/EV1000 versus standard practice. The sample size of 30 patients per group was calculated based on data from a previous study, an α value of 0.05, a β value of 0.2, and a 30% decrease in ICU stay. Sixty patients undergoing CABG with CPB at Srinagarind Hospital or Queen Sirikit Heart Center of the Northeast between July 2018 and June 2020 will be recruited. They will be divided into 2 groups: EV1000 and Control. The intraoperative hemodynamic optimization in the EV1000 was managed using goal-directed therapy via the FloTrac/EV1000 platform and the Control was managed using a standard protocol as described in the study of Tribuddharat et al. The extracted data for comparison were: demographic and clinical data, CVT ICU stay, ventilator time in CVT ICU, postoperative complications, and hospital stay. The ICU stay of both groups will be compared.

Assessing the daily CVT ICU cost

We will evaluate the ICU cost of the CVT ICU of Srinagarind Hospital by recruiting another group of patients who were admitted to the CVT ICU during October 2021 to identify the average daily cost. The cost of a FloTrac sensor and the ICU cost saved will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who underwent CABG with CPB.

Exclusion Criteria:

* Patients who required an intra-aortic balloon pump or extracorporeal membrane oxygenator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective CABG with CPB at Srinagarind Hospital or Queen Sirikit Heart Center of the Northeast between July 2018 and June 2020.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
ICU stay | 1 month
  The duration the patient was admitted in CVT ICU.

SECONDARY OUTCOMES:
Average daily ICU cost | 1 month
  The average cost per day of CVT ICU

CONTACTS AND LOCATIONS:
Overall Officials: Sirirat Tribuddharat, MD, PhD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Thepakorn Sathitkarnmanee, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tribuddharat S, Sathitkarnmanee T, Ngamsangsirisup K, Nongnuang K. Efficacy of Intraoperative Hemodynamic Optimization Using FloTrac/EV1000 Platform for Early Goal-Directed Therapy to Improve Postoperative Outcomes in Patients Undergoing Coronary Artery Bypass Graft with Cardiopulmonary Bypass: A Randomized Controlled Trial. Med Devices (Auckl). 2021 Jun 28;14:201-209. doi: 10.2147/MDER.S316033. eCollection 2021. PMID 34234581
- [Result] Tribuddharat S, Sathitkarnmanee T, Ngamsaengsirisup K, Sornpirom S. Efficacy of early goal-directed therapy using FloTrac/EV1000 to improve postoperative outcomes in patients undergoing off-pump coronary artery bypass surgery: a randomized controlled trial. J Cardiothorac Surg. 2022 Aug 21;17(1):196. doi: 10.1186/s13019-022-01933-4. PMID 35989328
- [Result] Aya HD, Cecconi M, Hamilton M, Rhodes A. Goal-directed therapy in cardiac surgery: a systematic review and meta-analysis. Br J Anaesth. 2013 Apr;110(4):510-7. doi: 10.1093/bja/aet020. Epub 2013 Feb 27. PMID 23447502
- [Result] Chong MA, Wang Y, Berbenetz NM, McConachie I. Does goal-directed haemodynamic and fluid therapy improve peri-operative outcomes?: A systematic review and meta-analysis. Eur J Anaesthesiol. 2018 Jul;35(7):469-483. doi: 10.1097/EJA.0000000000000778. PMID 29369117
- [Result] Gutierrez MC, Moore PG, Liu H. Goal-directed therapy in intraoperative fluid and hemodynamic management. J Biomed Res. 2013 Sep;27(5):357-65. doi: 10.7555/JBR.27.20120128. Epub 2013 Mar 10. PMID 24086168
- [Result] Neumann K, Muhr G, Breitfuss H. [Primary humerus head replacement in dislocated proximal humeral fracture. Indications, technique, results]. Orthopade. 1992 Apr;21(2):140-7. German. PMID 1594234
- [Result] Lefrant JY, Garrigues B, Pribil C, Bardoulat I, Courtial F, Maurel F, Bazin JE; CRREA Study Group; AzuRea Group. The daily cost of ICU patients: A micro-costing study in 23 French Intensive Care Units. Anaesth Crit Care Pain Med. 2015 Jun;34(3):151-7. doi: 10.1016/j.accpm.2014.09.004. Epub 2015 May 16. PMID 25986476